CLINICAL TRIAL: NCT00304473
Title: Fast Titration of Quetiapine Versus Conventional Titration in the Treatment of Schizophrenia/Schizoaffective Disorder: a Randomised, Parallel Group Open Trial
Brief Title: Fast Titration in the Treatment of Schizophrenia, Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1449C00001
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate

SUMMARY:
Assess the efficacy of a fast titration of quetiapine to the current titration approved by the regulatory authorities.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, at least 18 years old, inpatients with relapse Schizophrenia all subtypes, and with a CGI (Clinical Global Impression) score >=4.

Exclusion Criteria:

* Pregnancy or breast-feeding, patients treated with Clozapine within 28 days of randomization, patients with a known arrhythmia, any psychotic disorders not defined in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-08; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Compare the safety and tolerability of a fast titration of quetiapine to the current titration approved by the regulatory authorities.

SECONDARY OUTCOMES:
Assess the efficacy of a fast titration of quetiapine to the current titration approved by the regulatory authorities.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Taiwan Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Taoyuan District, Taiwan